CLINICAL TRIAL: NCT06378723
Title: Investigation of the Relationship Between Functionality, Trunk Control and Balance in Children With Cerebral Palsy
Brief Title: The Relationship Between Upper Extremity Functionality, Trunk Control and Balance in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Other Study IDs: 2024/01/24
Record Dates: First submitted 2024-02-14; First posted 2024-04-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Diplegic Cerebral Palsy; Balance; Distorted
Keywords: cerebral palsy; upper extremity; trunk control; functionality; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Children: Healthy children between the ages of 8 and 18 will be included in the study. Children with hearing and vision loss will be excluded from the study in order not to affect balance disorders.
  Interventions: Other: Balance Tests
- Cerebral Palsy Children: Cerebral Palsy children between the ages of 8 and 18 will be included in the study. Children with hearing and vision loss will be excluded from the study in order not to affect balance disorders. In order to standardize their mobility, those with Gross Motor Function Classification levels 1 and 2 will be included in the study.
  Interventions: Other: Balance Tests

INTERVENTIONS:
Other: Balance Tests — With the scales and tests the children trunk control, quality of upper extremity skills, single leg stance duration will be measured

SUMMARY:
The aim of this study is to examine the relationship between trunk control, upper extremity functionality and balance in children with cerebral palsy and to compare this relationship with healthy sedentary children.This study is carried out through Eastern Mediterranean University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Pediatric Rehabilitation Unit.

DETAILED DESCRIPTION:
23 children with Cerebral Palsy and 30 healthy children will be included in the study, and the families of all children participating in the study will sign an informed consent form.After signing the consent form from the families of the children included in the study, their demographic information will be recorded and their Gross Motor Function Classification System levels will be determined.

Children's upper extremity functionality will be evaluated with the Quality of Upper Extremity Skills Test. To determine their functional balance, the Single-Leg Stance Test and the Four Step Square Test are measured. Additionally, balances will be determined by the Trunk Control Measurement Scale. Evaluations are made using tables and chairs. Evaluations take approximately 60 minutes, depending on the condition of the children, and all evaluations will be made one-on-one by the physiotherapist. In the study where power analysis was performed, 50 child evaluations were deemed appropriate. Statistical Package for the Social Sciences package program is used to analyze the data. Whether the data complies with normal distribution will be evaluated using the Shapiro Wilk Test and histogram graphs. Descriptive statistics are given as mean, standard deviation, median, number and percentage. Numerical data between groups are compared using Student's t test and Mann Whitney U test. Categorical data will be compared using the Chi Square test. Spearman's correlation test was used for correlation analysis, p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8-18,
* Gross Motor Function Classification System level 1-2,
* Do not have severe visual or hearing impairment,
* Does not have any cooperation problems that would hinder communication,
* Children who have had Botulinum Toxin-A injection

Exclusion Criteria:

* Those with GMFC level 3-4-5,
* Children who had surgery within the last six months were not included in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cerebral Palsy and healthy children between the ages of 8 and 18 will be included in the study. Children with hearing and vision loss will be excluded from the study in order not to affect balance disorders. In order to standardize their mobility, those with GMFC levels 1 and 2 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
trunk control | one month
  All the children will be measured with the Trunk Control Measurement Scale. This test includes 15 items that measure static and dynamic sitting balance, two components of trunk control during functional activities. All items are scored on 2, 3 or 4 points and are administered bilaterally. The total score is between 0-58. A high score indicates good performance.
upper extremity functionality | one month
  All the children will be measured with the Quality of upper extremity skills test. This test evaluates the quality of upper extremity movements; It evaluates in 4 different areas: independent movements, grasping, weight bearing and protective extension. In protective extension, falling to the front, back and side using the arms is evaluated. A "yes" or "no" score is given depending on the completion of each action or task. Scores in these four areas are added together for a total score. Additionally, hand function, spasticity and cooperation are also evaluated. In hand function evaluation, 0 to 10 points are marked for the right hand, left hand and bilaterally. In cooperation, children's cooperation statuses are marked as "not cooperative", "partially cooperative" and "fully cooperative". During the evaluation, the child is not allowed to use any devices for the upper extremity. Both the child's right and left upper extremities are scored separately. Total score is between 0 and 100.
balance | one month
  all the children will be measured with the Four Step Square Test and Single leg Stance test. It is desirable to maintain this posture for as long as possible during the test. The test and duration begin with the foot being lifted off the ground. The test is repeated twice and the best time measured is noted in seconds (for single leg stance). The test begins with one foot of the individual touching the ground in the 2nd square and ends with the last foot touching the ground in the 1st square. The test is repeated twice for each individual and the test score completed in the shortest time is recorded in seconds (four step square test).
Weight and Height | one month
  Weight and height will be combined to report BMI in kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Emine Tuzun, Prof, Study Director — Eastern Mediterranean University
Locations (2):
- Eastern Mediterranean University, Famagusta, Cyprus
- Yeni Sihirli Eller Özel Eğitim ve Rehabilitasyon Merkezi, Adana, Çukurova, Turkey (Türkiye)